CLINICAL TRIAL: NCT07346885
Title: A Comparison of the Efficacy of Lumbar and Sacral Plexus Block Versus Fascia Iliaca Block Combined With Low-Dose Spinal Anesthesia in Patients Undergoing Surgery for a Femoral Neck Fracture
Brief Title: Lumbar-Sacral Plexus Block vs Fascia Iliaca Block Plus Low-Dose Spinal Anesthesia for Femoral Neck Fracture Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BursaYIEAH-2024 TBEK 2025/12-1
Record Dates: First submitted 2025-12-29; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Femoral Neck Fractures; Nerve Block
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbar and Sacral Plexus Block Group (Active Comparator): Patients will receive combined lumbar and sacral plexus blocks as the primary regional anesthesia technique for femoral neck fracture surgery, performed by the attending anesthesiologist according to institutional practice.
  Interventions: Procedure: Lumbar and Sacral Plexus Block
- Fascia Iliaca Block Combined with Low-Dose Spinal Anesthesia Group (Active Comparator): Patients will receive low-dose spinal anesthesia combined with a supra-inguinal fascia iliaca block for surgical anesthesia and postoperative analgesia.
  Interventions: Procedure: Fascia Iliaca Block Combined with Low-Dose Spinal Anesthesia

INTERVENTIONS:
Procedure: Lumbar and Sacral Plexus Block — For lumbar and sacral plexus blocks, a 10-15 cm ultrasound-visible peripheral nerve block needle and a nerve stimulator will be used. For lumbar plexus shamrock imaging and sacral plexus blocks, parasacral imaging will be used. 0.5% bupivacaine will be used as the local anesthetic.
  Arms: Lumbar and Sacral Plexus Block Group
Procedure: Fascia Iliaca Block Combined with Low-Dose Spinal Anesthesia — Spinal anesthesia will be administered using a 25-gauge Quincke needle. After positioning the patient on the side to be operated on in a lateral position, hypobaric spinal anesthesia will be administered through an appropriate (L3-4 or L4-5) with 1.5 cc of local anesthetic mixture. Before receiving spinal anesthesia, patients will undergo a supra-inguinal fascia iliaca block with 20 to 30 milliliters of 0.25% local anesthetic (bupivacaine).
  Arms: Fascia Iliaca Block Combined with Low-Dose Spinal Anesthesia Group

SUMMARY:
Femoral neck fracture surgery in elderly patients is frequently complicated by intraoperative hypotension and inadequate postoperative analgesia. Regional anesthesia techniques are increasingly preferred to reduce hemodynamic instability and improve pain control. This prospective observational study aims to compare the efficacy of lumbar and sacral plexus block with fascia iliaca block combined with low-dose spinal anesthesia in terms of severe intraoperative hypotension and postoperative analgesic outcomes in patients undergoing surgery for femoral neck fracture.

DETAILED DESCRIPTION:
The global incidence of hip fractures continues to rise, and most patients require surgical intervention. Due to advanced age, frailty, and multiple comorbidities, anesthetic management in this population is particularly challenging. Intraoperative hypotension has been shown to be associated with increased short- and long-term mortality, regardless of the anesthetic technique used.

To reduce the incidence of hypotension, various neuraxial and peripheral nerve block techniques have been investigated. While spinal anesthesia provides reliable surgical conditions, it may still cause significant hypotension. Peripheral nerve blocks, such as lumbar and sacral plexus blocks or fascia iliaca block, tend to preserve hemodynamic stability and are associated with a lower incidence of motor blockade.

Recently, combined techniques using low-dose spinal anesthesia together with fascial plane blocks have been introduced to balance the advantages of neuraxial anesthesia and peripheral nerve blocks. However, there is still no consensus on the optimal regional anesthesia strategy to minimize severe hypotension while ensuring effective analgesia in patients undergoing femoral neck fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

->18 years and <90 years

* American Society of Anesthesiologists score between I and IV
* Patients who will undergo femoral neck fracture surgery

Exclusion Criteria:

* Previous local anesthetic allergy
* Those with bleeding diathesis disorder
* Having a mental disorder
* Those who are allergic to the drugs used
* Patients who did not consent to participate in the study
* Presence of infection in the block area
* Body mass index >30
* Preoperative or intraoperative general anesthesia
* Patients for whom consent cannot be obtained
* Pregnant patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Severe Intraoperative Hypotension | Intraoperative period
  Severe hypotension defined as mean arterial pressure (MAP) < 65 mmHg lasting longer than 12 minutes during surgery

SECONDARY OUTCOMES:
intraoperative haemodynamic parameters | intraoperative 2 hours
  non-invasive systolic, diastolic and mean arterial pressure
  mean arterial pressure (mm/hg)
Total Intraoperative Sedative and Analgesic Drug Consumption | intraoperative 2 hours
  Total intraoperative sedative and analgesic drug consumption will be recorded, including the cumulative dose of sedative agents (e.g., propofol, midazolam) and analgesic agents (e.g., fentanyl or equivalent opioids) administered during surgery.
Estimated Intraoperative Blood Loss (mL) | intraoperative 2 hours
  Estimated intraoperative blood loss will be assessed by the anesthesiology team based on suction canister volume minus irrigation fluids and surgical sponge weight estimation, as routinely used in clinical practice.
Postoperative Pain Intensity Assessed by the Numeric Rating Scale (NRS) | postoperative 24 hour
  Pain intensity will be assessed using the Numeric Rating Scale (NRS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Pain scores will be recorded at rest and during movement
Intraoperative Vasopressor Consumption | Intraoperative period
  Total dose of vasopressors administered
Length of Hospital Stay (days) | From the day of surgery through hospital discharge (up to 30 days)
  Length of hospital stay will be defined as the number of days from the day of surgery until hospital discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences,,Bursa Yuksek Ihtisas Training and Research Hospital,, Bursa, Turkey (Türkiye)